CLINICAL TRIAL: NCT02678845
Title: Project Collabri. The Effect of a Collaborative Care Model for Treatment of Depression in Primary Care in Denmark - A Cluster Randomized Clinical Superiority Trial
Brief Title: Project Collabri for Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2013-203-D
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment according to the Collabri model (Experimental): Participants in this group will recive treatment according to the Collabri model which is a Danish model for collaborative care between primary and secondary care for depression, social phobia, generalized anxiety and panic disorder
  Interventions: Other: Treatment according to the Collabri model
- Treatment as usual (No Intervention): Control group. Participants in this group will recive treatment as usual. This means that participants will recive treatment corresponding to what their GP normally would offer as treatment. E.g. this could be refferal to a psychologist or psychiatrist and/or medicine.

INTERVENTIONS:
Other: Treatment according to the Collabri model — The Collabri Model is a complex intervention and consists of a number of treatment modalities. The Collabri Model includes the following elements: A multi-professional approach to treatment including a care manager, scheduled monitoring and review, enhanced inter-professional communication and a structured treatment plan. It further integrates: Recruitment of staff with psychiatric experience, training of general practitioner and care manager, use of instruments for detection and follow-up, education and treatment of the patient, supervision from a psychiatric specialist, guided self-help, patient- and relative involvement and a stepped care approach to treatment where treatment is always commenced on the least invasive and least resource-demanding level.
  Arms: Treatment according to the Collabri model

SUMMARY:
The purpose of this study is to determine whether treatment of patients with depression according to the Collabri Model is more effective in reducing symptoms compared to treatment as usual (TAU)

DETAILED DESCRIPTION:
Background:

Depression is a common disease mostly treated in general practice. Diagnose and evidence based treatment in general practice today is not optimal (e.g. lack of continuity in disease management and lack of treatment opportunities).

International studies show effect of collaborative care on depression, but is not directly applicable into a Danish context.

A Danish model for collaborative care treatment of people with depression, generalized anxiety disorder, social phobia and panic disorder (the Collabri Model) is developed. The Collabri model consists of a multi-professional approach to treatment, scheduled monitoring and review, enhanced inter-professional communication and a structured treatment plan.

Objectives:

to investigate the effect of the Collabri model for depression and further investigate two methods for detection of depression; standard detection and case finding.

Methods:

Two researcher-blinded cluster-randomized controlled studies with an intervention group (treatment according to the Collabri model) and a control group (TAU). Participants are 480 patients with depression consulting their general practitioner.

Results:

Primary outcome for the collaborative care study on depression is depression symptoms, measured with BDI at 6 months.

Discussion:

The results will contribute new knowledge on collaborative care for depression and anxiety in Danish conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18+ years
* Danish speaking
* Diagnosis of current depression using the Mini International Neuropsychiatric Interview (MINI) (DSM IV) by researchers that have been trained in using MINI and according to the ICD-10 criteria or when diagnosed by GP after conference with a psychiatrist in Project Collabri
* The patient has given her/his written informed consent to participate in the trial at the described terms

Exclusion Criteria:

* High risk of suicide assessed in the Mini International Neuropsychiatric Interview (MINI) and/or by general practitioner
* Psychotic condition detected in the MINI and/or by general practitioner
* Patients with a diagnosis of dementia
* Pregnancy
* Alcohol or substance misuse that hinders the person participating in Collabri treatment as assessed by the practitioner or researcher at inclusion interview
* Patients that are in current psychological or psychiatric treatment due to anxiety or depression
* Patients with a pending disability pension case
* Patients who have been treated for anxiety or depression within the last 6 months
* For patients in the intervention group: Patients with depression who wants treatment cf. the Danish psychologist scheme and do not want the reference to the psychologist preceded by other treatment, cf. the Collabri model
* For patients in the intervention group: If the patient at the first point of contact with the general practitioner after inclusion by a research assistant is referred to treatment as a part of the secondary psychiatric care system.
* Patients who are assessed by the general practitioner as medically unstable making it impossible for the patient to adhere to treatment
* OCD, PTSD, bipolar affective disorder as assessed in the MINI and/or by the general practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Degree of depression measured by the Beck Depression Inventory (BDI) | At 6 months follow up after baseline
  The measure is self-reported

SECONDARY OUTCOMES:
Degree of anxiety measured by the Beck Anxiety Inventory (BAI) | At 6 months follow up after baseline
  The measure is self-reported
Psychological stress measured with the Symptom Checklist (SCL-92) | At 6 months follow up after baseline
  The measure is self-reported
Functional impairment measured with the Global Assessment of Functioning (GAF-F split version) | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview

OTHER OUTCOMES:
Degree of depression measured by the Beck Depression Inventory (BDI) | At 15 months follow up after baseline
  The measure is self-reported
Degree of anxiety measured by the Beck Anxiety Inventory (BAI) | At 15 months follow up after baseline
  The measure is self-reported
Psychological stress measured with the Symptom Checklist (SCL-92) | At 15 months follow up after baseline
  The measure is self-reported
Functional impairment measured with the Global Assessment of Functioning (GAF-F split version) | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview
Quality of life measured with the WHO-5 | At 6 months follow up after baseline
  The measure is self-reported
Quality of life measured with the WHO-5 scale | At 15 months follow up after baseline
  The measure is self-reported
Personal and social performance measured with the Personal and Social Performance scale (PSP) | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview
Personal and social performance measured with the Personal and Social Performance scale (PSP) | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview
Side effects measured by the PRISE questionnaire | At 6 months follow up after baseline
  The measure is self-reported
Side effects measured by the PRISE questionnaire | At 15 months follow up after baseline
  The measure is self-reported
Health-related quality of life measured with the EQ-5D | At 6 months follow up after baseline
  The measure is self-reported
Health-related quality of life measured with the EQ-5D | At 15 months follow up after baseline
  The measure is self-reported
Functional impairment measured with Sheehan Disability Scale (SDS) | At 6 months follow up after baseline
  The measure is self-reported
Functional impairment measured with Sheehan Disability Scale (SDS) | At 15 months follow up after baseline
  The measure is self-reported
Sick leave | At 6 months follow up after baseline
  The measure is obtained from the Danish DREAM database
Sick leave | At 15 months follow up after baseline
  The measure is obtained from the Danish DREAM database
Self-efficacy measured with the subscale "Obtain Help from Community, Family, Friends" from the Chronic Disease Self-Efficacy Scale | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Obtain Help from Community, Family, Friends" from the Chronic Disease Self-Efficacy Scale | At 15 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Control/Manage Depression Scale" from the Chronic Disease Self-Efficacy Scale | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Control/Manage Depression Scale" from the Chronic Disease Self-Efficacy Scale | At 15 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Personal Control" from The Revised Illness Perception Questionnaire (IPQ-R) | At 6 months follow up after baseline
  The measure is self-reported
Self-efficacy measured with the subscale "Personal Control" from The Revised Illness Perception Questionnaire (IPQ-R) | At 15 months follow up after baseline
  The measure is self-reported
Apathia | At 6 months follow up after baseline
  The measure is obtained through a semi-structured interview
Apathia | At 15 months follow up after baseline
  The measure is obtained through a semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD PhD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brinck-Claussen UO, Curth NK, Christensen KS, Davidsen AS, Mikkelsen JH, Lau ME, Lundsteen M, Csillag C, Hjorthoj C, Nordentoft M, Eplov LF. Improving the precision of depression diagnosis in general practice: a cluster-randomized trial. BMC Fam Pract. 2021 May 7;22(1):88. doi: 10.1186/s12875-021-01432-w. PMID 33962564
- [Derived] Curth NK, Brinck-Claussen UO, Hjorthoj C, Davidsen AS, Mikkelsen JH, Lau ME, Lundsteen M, Csillag C, Christensen KS, Jakobsen M, Bojesen AB, Nordentoft M, Eplov LF. Collaborative care for depression and anxiety disorders: results and lessons learned from the Danish cluster-randomized Collabri trials. BMC Fam Pract. 2020 Nov 18;21(1):234. doi: 10.1186/s12875-020-01299-3. PMID 33203365
- [Derived] Brinck-Claussen UO, Curth NK, Davidsen AS, Mikkelsen JH, Lau ME, Lundsteen M, Csillag C, Christensen KS, Hjorthoj C, Nordentoft M, Eplov LF. Collaborative care for depression in general practice: study protocol for a randomised controlled trial. Trials. 2017 Jul 21;18(1):344. doi: 10.1186/s13063-017-2064-7. PMID 28732523